CLINICAL TRIAL: NCT05917496
Title: Analysis of Parental Support in Families Using the LENA After Early Cochlear Implantation
Acronym: ACLEIC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230423; 2023-A00405-40 (Other: IDRCB Number)
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Profound Congenital Deafness; Cochlear Implantation
Keywords: Profound congenital deafness; Early cochlear implantation; Language environment; Child's language development; Speech therapy assessment; Language ENvironment Analysis (LENA) tool

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Children aged 11 months to 21 months on the day of inclusion in the study, with profound congenital deafness and having benefited from unilateral or bilateral cochlear implantation before 18 months of life inclusive, followed at Necker-Enfants Malades hospital and who receive a speech therapy.
  Interventions: Other: LENA tool: Language ENvironment Analysis; Behavioral: Return of the analysis of the data of LENA

INTERVENTIONS:
Other: LENA tool: Language ENvironment Analysis — Recording of the language environment of the child at home, in daily environment, with the LENA.
  The parameters recorded relate to four domains: "adult words", "conversation turns", "child vocalizations" and "exposure to electronic media".
  The LENA box is worn for 10-16 hours, with a minimum of 10 consecutive hours. the families make 2 separate recordings of 6 months at T1 and T2.
Behavioral: Return of the analysis of the data of LENA — The analysis of the LENA data is carried out by the speech therapist using the LENA Pro Version Software v3.4, during the times T1 and T2. The return of the analysis of the data collected via the LENA will be made to the family of the patient after T1 and after T2 and personalized advice will then be given to parents with the aim of improving their child's language skills.

SUMMARY:
The language environment that influences the child's language development has been studied using different subjective tools, mainly audio and/or video recording and manual transcriptions. The linguistic results of the implanted deaf child are dependent on the age at the implant, but also on the auditory and linguistic stimulation in the first months following the placement of the implant. Parents are the main actors in the child's language development. Professionals can rely on the LENA tool: Language ENvironment Analysis, which objectifies the language environment of the child at home in his daily environment. It is possible to obtain statistics on the number of adult words received by the child, the number of words produced by the child as well as the exposure to media and noise. On the basis of this quantitative data, the family can be supported in an attempt to optimize the conditions for receiving their child's speech.

The purpose of this study is to analyze the effect of speech therapy parental support using the data provided by the Language ENvironment Analysis (LENA) tool, in a pediatric population implanted early, i.e. before the age of 18 months and aged under 24 months inclusive at the start of their participation in the study.

DETAILED DESCRIPTION:
The language environment that influences the child's language development has been studied using different subjective tools, mainly audio and/or video recording and manual transcriptions. The linguistic results of the implanted deaf child are dependent on the age at the implant, but also on the auditory and linguistic stimulation in the first months following the placement of the implant. Parents are the main actors in the child's language development. Professionals can rely on the LENA tool: Language ENvironment Analysis, which objectifies the language environment of the child at home in daily environment. On the basis of this quantitative data provided by the LENA, the family can be supported in an attempt to optimize the conditions for receiving their child's speech.

The purpose of this study is to analyze the effect of speech therapy parental support using the data provided by the Language ENvironment Analysis (LENA) tool, in a pediatric population implanted early, i.e. before the age of 18 months and aged under 24 months inclusive at the start of their participation in the study.

The LENA tool was validated in French version in 2015. It is a system of recording and automatic analysis of the language environment of the child using a box worn for 10-16 hours, with a minimum of 10 consecutive hours. For the study, the families make 2 separate recordings of 6 months at home (T1 and T2) then, a centralized analysis of all the data is carried out by the speech therapist using adapted software, the LENA Pro Version Software v3.4, during the times T1 and T2. The return of the analysis of the data collected via the LENA will be made to the family after T1 and after T2.

The parameters resulting from this analysis relate to four domains: "adult words", "conversation turns", "child vocalizations" and "exposure to electronic media". Average numerical scores expressed in percentiles are published at the end of the analysis. Individual scores are then compared to a standard expressed as percentiles. The content of the conversations will not be listened to and only numerical scores will be used for each of the parameters studied and obtained by computer analysis.

ELIGIBILITY:
Inclusion Criteria:

* Have profound congenital deafness
* Have been implanted between 8 months and 18 months
* Have had a unilateral or bilateral cochlear implant for 3 months
* Be between 11 months and 21 months old on the day of inclusion
* Constant wearing of the implant
* Benefit from speech therapy
* Have a French-speaking parent
* Information and non-opposition of holders of parental authority to participate in the study

Exclusion Criteria:

* Syndromic deafness or auditory nerve aplasia
* Micro-cochlea or partial insertion of the electrode bundle
* CHARGE syndrome (acronym for Coloboma, Heart defect, Atresia choanae, Retarded growth and development, Genital hypoplasia, Ear anomalies/deafness or in French coloboma, cardiac malformation, choanal atresia, growth retardation and/or mental retardation, genital hypoplasia, ear abnormalities/deafness)
* Deafness with significant central involvement (cytomegalovirus, meningitis)
* Proven major disorders that can impact language development (Autism Spectrum Disorder, mental retardation, etc.)
* Non-daily wearing of the cochlear implant
* Proven uncorrected visual disturbances interfering with the performance of language level assessment tests

Ages: 11 Months to 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 24 months with profound congenital deafness and having benefited from unilateral or bilateral cochlear implantation before 18 months of life inclusive, followed at Hôpital Necker-Enfants Maladies and who receive a speech therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of conversation turns | 6 months
  Comparison of the variation in language environment for the number of conversation turns recorded at T1 and the number of conversation turns recorded at T2 after speech therapy support offered at T1 and based on data provided by the Language ENvironment Analysis (LENA) tool.
  Average numerical scores expressed in percentiles are produced at the end of the analysis. The individual scores are then compared with a standard expressed in percentiles.
Receptive lexical level | 6 months
  Receptive lexical level measured by the speech therapy test (IFDC, French inventories of Communicative Development) at T1 and T2.
  Each child's individual result is given in percentiles according to chronological age. It is based on an evaluation sheet with benchmarks in percentiles (10th to 90th) or percentages.
Correlation between the number of conversation turns parameter and the receptive lexical level | 6 months
  The correlation between the "conversation turns" parameter recorded at T1 and T2 and the receptive lexical level measured by the speech therapy test (IFDC, French inventories of Communicative Development) at T1 and T2 will be carried out.

SECONDARY OUTCOMES:
Link between 3 language environment parameters: adult words, child vocalization, exposure to electronic media and the receptive lexical level | 6 months
  To study the link between the 3 others language environment parameters (adult words, child vocalization, exposure to electronic media), evaluated by the LENA system and the receptive lexical level, measured by the standardized speech therapy test carried out at T1 and T2.
  Average numerical scores expressed in percentiles are produced at the end of the analysis. The individual scores are then compared with a standard expressed in percentiles.
Acceptability of the use of the LENA tool for children under 3 years | 24 months
  Evaluate the acceptability of the use of the LENA tool for children under 3 years old implanted between 8 and 18 months using the acceptability questionnaire completed by the parents concerning the use of the LENA system in their child at T1 and T2.
  An "acceptability" score will be calculated on the basis of this questionnaire and expressed as a percentage: the questionnaire consists of 6 questions, each answer worth 2, 1 or 0 points (i.e. a maximum gross score of 12 points), then the gross score divided by 6 and multiplied by 50 to obtain a percentage score (100% corresponding to excellent acceptability).
Protocolizing the individual strategies given to help and support parents to enrich their child's language environment | 6 months
  Analyze the individual results obtained from the language environment data collected from the LENA tool, in order to provide personalized advice to parents after T1 and T2, with the aim of improving their child's language environment. Comparison of individual scores at T1 and T2 for the 4 parameters evaluated by the LENA system ("adult words", "conversation turns", "child vocalizations" and "exposure to electronic media") with the means scores obtained. Carry out a process of protocolizing the individual strategies given to help and support parents in enriching their child's language environment.
Family participation during speech therapy | 6 months
  Comparison of scores from the family participation scale at T1 and T2. The speech and language therapist subjectively assesses the family's involvement by assigning a number corresponding to the level of involvement and motivation: the calibration is made from 1 (limited involvement) to 5 (ideal involvement).

CONTACTS AND LOCATIONS:
Overall Officials: Clara LEGENDRE, speech therapist, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Natalie LOUNDON, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrose SE, VanDam M, Moeller MP. Linguistic input, electronic media, and communication outcomes of toddlers with hearing loss. Ear Hear. 2014 Mar-Apr;35(2):139-47. doi: 10.1097/AUD.0b013e3182a76768. PMID 24441740
- [Background] Canault M, Le Normand MT, Foudil S, Loundon N, Thai-Van H. Reliability of the Language ENvironment Analysis system (LENA) in European French. Behav Res Methods. 2016 Sep;48(3):1109-24. doi: 10.3758/s13428-015-0634-8. PMID 26174716
- [Background] Canault, M., Le Normand, M.-T., & Thai Van, H. (2017). LENATM (Language ENvironment Analysis System) : Un système de reconnaissance automatique de la parole et de l'environnement langagier de l'enfant. Enfance, 2(2), 199 216. https://doi.org/10.3917/enf1.172.0199
- [Background] Coquet, F., Roustit, J. (2009).Batterie EVALO 2-6 : un nouvel outil d'EVAluation du développement du Langage Oral chez l'enfant de 2 ans 3 mois à 6 ans 3 mois. UPLF Infos, janvier. Union Professionnelle des Logopèdes Francophones. Belgique
- [Background] Dunn LM., Theriault-Whalen CM., Dunn LM. (1993). Echelle de Vocabulaire en Images Peabody. (EVIP). Toronto (Canada) : Psychan.
- [Background] Gilkerson J. & Richards J. A. (2009) The power of talk: Impact of adult talk, conversational turns, and TV during the critical 0-4 years of child development (Technical Report LTR-01-2). Retrieved from: http://www.lenababy.com/pdf/The_Power_of_Talk.pdf
- [Background] Fenson L., Dale P., Reznick S., Thal D., Bates E., Hartung J., Tethick S., Reilly J. : MacArthur Communicative Development Inventories : User's guide and technical manual, San Diego, CA, Singular Publishing Group, 1993.
- [Background] Hart B. & Risley T. (1995). Meaningful differences in the everyday experience of young American children. Baltimore: Brookes.
- [Background] Haute Autorité de Santé. (2009, décembre). Recommandations de bonne pratique : surdité de l'enfant : accompagnement des familles et suivi de l'enfant de 0 à 6 ans, hors accompagnement scolaire. HYPE://www.has-sante.fr/jcms/c_922867/fr/surdite-de-l-enfant-accompagnement-des- familles-et-suivi-de-l-enfant-de-0-a-6-ans-hors-accompagnement-scolaire
- [Background] Moeller MP. Early intervention and language development in children who are deaf and hard of hearing. Pediatrics. 2000 Sep;106(3):E43. doi: 10.1542/peds.106.3.e43. PMID 10969127
- [Background] Moeller MP, Carr G, Seaver L, Stredler-Brown A, Holzinger D. Best practices in family-centered early intervention for children who are deaf or hard of hearing: an international consensus statement. J Deaf Stud Deaf Educ. 2013 Oct;18(4):429-45. doi: 10.1093/deafed/ent034. PMID 24030911
- [Background] Kern, S. & Gayraud, G., 2010,